CLINICAL TRIAL: NCT00951353
Title: Immune Development and Alloimmunity in Pediatric Renal Transplant Recipients
Brief Title: Immune Development in Pediatric Transplantation (IMPACT)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-02
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Chronic Kidney Failure; End Stage Renal Disease
Keywords: Transplantation; Kidney Failure; End Stage Renal Disease; Pediatric
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Renal Transplant Recipients

SUMMARY:
Transplantation is the preferred method of treatment for end-stage renal disease (ESRD) in children. Over the past forty years, the use of newer immunosuppressive drugs has decreased the risk for organ rejection considerably, and improved short-term outcomes. However, these costly and complicated life-long treatment regimens also cause serious side effects. This has been particularly true for children, who undergo treatment with these drugs at the same time they are transitioning, physically and emotionally, from childhood to adulthood. These factors lead to significantly reduced life-spans, decreased drug regimen adherence, and an increased need for re-transplantation, as compared with adults.

Current immunosuppressive procedures and strategies for children mimic those for adults, despite the difference between the two populations' immune systems and needs. New strategies aimed at tailoring to an individual child's needs would both reduce the risk of complications and improve outcomes. The purpose of this study is to generate information which will help to change the current practice of pediatric transplantation into one that is more individualized and preventative.

DETAILED DESCRIPTION:
Over the past forty years, the use of increasingly effective immunosuppressive drugs has decreased the risk for organ rejection (acute rejection, AR) considerably, and improved short-term outcomes. However, these costly and complicated life-long treatment regimens also cause serious complications in the long-term.

While transplant recipients live significantly longer lives than patients on dialysis, transplant recipients still have much shorter life spans than their healthy counterparts. Among reasons for this difference in life-expectancy are the immunosuppressive-drug related side effects that can lead to complications such as life threatening infections, malignancies, high blood pressure, heart disease, and diabetes. Additionally, certain drugs used to prevent organ rejection are known to contribute to renal damage, leading many patients to experience graft loss within 15 years. To that end, many children undergoing successful kidney transplantation require re-transplantation as adults. Therefore, while transplantation yields high success rates in the short-term, the drugs that are responsible for this early and temporary success are also the cause of later, serious complications. This is especially true for children, who endure extended drug exposures.

The purpose of this study is to explore the impact of viral exposure on children who receive immunosuppressive medications after renal transplantation; study the cellular changes associated with these influences; monitor medication adherence; and observe how all these factors affect the outcome of kidney transplantation in children. The hope is to better understand these processes to optimize future transplant therapies for the pediatric transplant recipient.

This study is designed to observe the immune system response during the first year after kidney transplant. Cells of the immune system in the recipient's blood, urine, and transplanted kidney will be tested to observe how the drugs used to prevent rejection influence them, if these cells change over time, and if they are related to kidney rejection. The comparisons will allow researchers to study how the developing immune system interacts with the kidney transplant. Blood from the kidney donor will be requested so that researchers can study how the recipient's immune system interacts with donor cells.

This study will also look closely at how well participants take prescribed medications. Since transplant medications are known to change the immune system, tests of the immune system cells will be compared to tests designed to measure how accurately medications are taken. Medication adherence will be measured using electronic medication bottle cap records, paper survey results, and drug levels in the blood. In this way, the study team hopes to learn about the impact of children's medications on their immune system.

This study will take place at multiple transplant centers in the United States. It is observational and will involve approximately 75 pediatric renal participants. The study will last for a total of 3 years, which includes a 2 year accrual period and 12 month follow up. Clinical treatment will be determined by standard of care at each participating center. There will be Baseline assessments which will occur before and on the day of transplantation and follow-up study visits will take place at months 1, 3, 6, 9, and 12 after transplant. Study assessments and specimens will also be collected at the time of each clinically indicated biopsy. Study assessments during these follow-up visits will include vital signs; review of current medications; questions related to adverse events (infection, rejection, graft failure, malignancy); treatment adherence surveys; and specimen collection for local and central laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian willing to provide informed consent, if necessary
* 1 to 20 years of age (before 21st birthday) at the time of enrollment
* Undergoing renal transplantation

Exclusion Criteria:

* Need for multi-organ transplantation
* Any prior history of organ transplantation
* Inability or unwillingness of participant of their legal guardian to give written informed consent or comply with study protocol

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric end-stage renal disease patients needing a kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy proven and treated (steroid pulse, taper, immunosuppressant medication changes) acute rejection Banff grade borderline or higher | 6 months after transplant

SECONDARY OUTCOMES:
Incidence of treated, clinically suspected rejection without biopsy | Throughout study
Incidence of biopsy proven and clinically relevant chronic allograft nephropathy | Throughout study
Incidence of infection and malignancy | Throughout study
Incidence of medication non-adherence in pediatric kidney transplant recipients using self report questionnaires and electronic monitoring bottle caps | Throughout study
Clinical impact of medication non-adherence with regard to the incidence of acute and chronic rejection | Throughout study
The degree to which a child's T Cells are predominately naïve, TEM, TCM, or TTM as measured by MFC | Throughout study
The heterologous alloreactivity of defined viral T cells for donor and third party alloantigens using MHC tetramers with specificity for CMV and EBV | Throughout study
The peripheral blood, urine, and allograft transcriptional phenotypes specific to the MFC-defined T cell phenotype | Throughout study
Formation of anti-donor HLA, non HLA, and MICA antibodies after transplantation as measured using Luminex platforms and microarray | Throughout study
Identification of specific proteins in blood and allograft as correlated with rejection | Throughout study
Barriers to adherence as indicated by AMBS, PMBS, and BMQ questionnaires | Throughout study
Candidate surrogate markers of immunosuppressive medication non-adherence: • Tacrolimus drug level variation • De novo immune activation using real time PCR message for perforin and granzyme B, and • Anti-HLA antibodies | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Allan D. Kirk, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - University of California at Los Angeles/ Mattel Children's Hospital, Los Angeles, California
  - Stanford University Medical Center/ Lucille Packard Children's Hospital, Palo Alto, California
  - Emory University/ Children's Healthcare of Atlanta, Atlanta, Georgia

REFERENCES:
- [Result] Ettenger R, Chin H, Kesler K, Bridges N, Grimm P, Reed EF, Sarwal M, Sibley R, Tsai E, Warshaw B, Kirk AD. Relationship Among Viremia/Viral Infection, Alloimmunity, and Nutritional Parameters in the First Year After Pediatric Kidney Transplantation. Am J Transplant. 2017 Jun;17(6):1549-1562. doi: 10.1111/ajt.14169. Epub 2017 Feb 1. PMID 27989013
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) program website — http://ctotc.org/
- Available data/document: Study Protocol: SDY951 — http://www.immport.org/immport-open/public/home/studySearch — ImmPort study identifier is SDY951.
- Available data/document: Complete set of descriptive data and results: SDY951 — http://www.immport.org/immport-open/public/home/studySearch — ImmPort study identifier is SDY951. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. This archive is in support of the NIH mission to share data with the public.